CLINICAL TRIAL: NCT02162225
Title: Phase 2 Study of Effects of Plasma Nitrite in Sickle Cell Anemia
Brief Title: Study of Beet Juice for Patients With Sickle Cell Anemia
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Enrollment was very slow. Hope to reopen as multi-site study
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: Wake Forest University (Other); National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Wake-58091; R37HL058091 (NIH)
Record Dates: First submitted 2014-06-09; First posted 2014-06-12 (Estimated); Last update posted 2018-08-02 (Actual); Status verified 2018-07

CONDITIONS: Sickle Cell Anemia
Keywords: Erythrocyte Deformability; Platelet Activation; Platelet Aggregation; Nitrite; Sickle Cell Anemia; Diet Therapy
MeSH Terms: conditions — Anemia, Sickle Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Beet Juice (Experimental): Volunteers will drink a single 8 ounce bottle of beet juice (Unbeetable) per day for 28 days.
  On days 1,14, and 28, the juice will be drunk just prior to having blood drawn. Blood will also be drawn 1.5 hours after drinking the juice on days 1,14, and 28.
  Interventions: Drug: beet juice (Unbeetable)

INTERVENTIONS:
Drug: beet juice (Unbeetable) — Volunteers will drink a single 8 ounce bottle of beet juice (Unbeetable) per day for 28 days.
  On days 1,14, and 28, the juice will be drunk just prior to having blood drawn. Blood will also be drawn 1.5 hours after drinking the juice on days 1,14, and 28.

SUMMARY:
The investigators hypothesize that increasing plasma nitrite using dietary nitrate will improve platelet function and red cell deformability and decrease MCHC in patients with sickle cell disease. The investigators will test this hypothesis through administration of daily intake of beetroot juice (Unbeetable - Performance Drink) to patients with sickle cell disease for 28 days. The investigators will evaluate the safety of daily beet root juice intake in patients with sickle cell disease. In addition, the investigators will measure MCHC, red cell deformability, and platelet function (activation and aggregation) in response to daily intake of beet root juice in this patient population.

DETAILED DESCRIPTION:
Sickle cell disease is caused by dysfunction of a mutant form of hemoglobin which polymerizes under hypoxic conditions, sickling the red blood cell. Sickling makes the cells rigid which contributes to vascular occlusion and much morbidity and mortality. Cycles of sickling and unsickling leads to calcium (Ca) influx which activates the gardos channel which pumps out potassium from the cells. Loss of potassium leads to dehydration, poor deformability, and increased mean corpuscular hemoglobin concentration (MCHC) in red blood cells. Increased MCHC leads to increased polymerization. Thus, a significant therapeutic goal for sickle cell disease has been to decrease MCHC by blocking the Ca-influx induced dehydration.

Rifkind and coworkers have shown that the NO+ donor sodium nitrosoprusside (SNP) can block Ca-induced loss of deformability when normal red blood cells are exposed to Ca and a Ca ionophore. The investigators have preliminary data showing that both NO activity donors SNP and nitrite can partially relieve loss of deformability due to cycles of sickling and unsickling in red cells from patients with sickle cell disease.

Low nitric oxide (NO) bioavailabilty secondary to red cell hemolysis has been proposed to contribute to pathology in sickle cell disease. Low NO could lead to poor protection against Ca-induced potassium loss described above. Another consequence of low NO is likely to be increased platelet activation; sickle cell disease is pro-thrombotic disease. NO reduces platelet aggregation and activation. It has been shown that an acute dietary nitrate intervention can reduce platelet aggregation in healthy volunteers. Nitrate is converted to nitrite which is converted to NO in the body.6 Improved platelet function is likely due to increasing NO bioavailability through the nitrate intervention.

In this pilot study, the safety of Beet Juice intake in patients with sickle cell disease will be evaluated using a self-administered health survey. Physiological effects of the Beet Juice will also be examined and the investigators hypothesize that increasing plasma nitrite using dietary nitrate will improve platelet function and red cell deformability and decrease MCHC in patients with sickle cell disease. The investigators will test this hypothesis through administration of daily intake of Beet Juice to patients with sickle cell disease for 28 days. The investigators will measure MCHC, red cell deformability, and platelet function (activation and aggregation) in response to the intervention.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of sickle cell anemia (Hb S/S or Hb S/beta thal0)
* no acute illness at the time of obtaining the study
* willingness to adhere to the study preparatory procedures including drinking the beet juice product daily
* willingness to give consent in order to participate

Exclusion Criteria:

* less than 19 years in age or older than 65
* smoke or chew tobacco
* currently take medications that affect stomach pH
* atrophic gastritis
* hypo-or hyperthyroidism
* Type I or II diabetes
* history of gout, kidney stones or hypotension
* pregnant
* aversion to the study-related testing procedures
* allergy, sensitivity or aversion to the study beetroot juice beverage
* suffered an acute sickle cell episode (involving hospitalization or a visit to the emergency room) within the past six months

Ages: 19 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2014-09; Primary Completion 2019-02 (Estimated); Study Completion 2019-04 (Estimated)

PRIMARY OUTCOMES:
Total Number of Participants with Adverse Events as a Measure of Safety and Tolerability as a function of time | up to 58 Days
  Physical symptoms will be assessed either by telephone or in person

SECONDARY OUTCOMES:
Changes in Red blood cell properties as a function of time | Days 1, 14, 28
  Blood will be drawn and used to measure red blood cell deformability and mean corpuscular hemoglobin concentration
Changes in Platelet function as a function of time | Days 1, 14, 28
  Blood will be drawn and used to measure platelets activation and aggregation

CONTACTS AND LOCATIONS:
Overall Officials: Natalia Dixon, MD, Principal Investigator — Wake Forest University Health Sciences; Daniel B Kim-Shapiro, PhD, Study Director — Wake Forest University
Locations (1):
- Wake Forest University School of Medicine, Winston-Salem, North Carolina, United States